CLINICAL TRIAL: NCT04605614
Title: A Phase I Study of 64Cu Pembrolizumab PET Imaging for In Vivo Expression of PD1
Brief Title: 64Cu-DOTA-pembrolizumab PET for the Study of PD1 Expression
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accruals
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080; NCI-2020-07955 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20080 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — pembrolizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, 64Cu-DOTA-pembrolizumab, PET) (Experimental): Patients receive pembrolizumab IV over 30 minutes, and within 6 hours also receive 64Cu-DOTA-pembrolizumab via slow IV push over > 1 minute on day 0. Patients then undergo PET over 60 minutes on day 1.
  Interventions: Radiation: Copper Cu 64-DOTA-pembrolizumab; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Radiation: Copper Cu 64-DOTA-pembrolizumab — Given IV
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial evaluates the best dose and side effects of copper (64Cu)-DOTA-pembrolizumab positron emission tomography (PET) for the study of PD1 expression. 64Cu is a radiotracer that binds to a molecule, PD1, that is found on immune cells that are found in the tumor. PD1 is short for 'programmed cell death protein 1'. When 64Cu-DOTA-pembrolizumab is injected into the patient's bloodstream, the 64Cu-pembrolizumab travels throughout the body and sticks to any tumor that has PD1 positive immune cells. Identifying the expression of PD1 in the tumor may help assess whether patients will respond to immunotherapy, and may detect clusters of immune cells when they are still too small to be detected by other Food and Drug Administration (FDA) approved techniques.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety and tolerability of unlabeled pembrolizumab followed by 64Cu-tetraxetan (DOTA)-pembrolizumab positron emission tomography, at each dose level, by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

SECONDARY OBJECTIVES:

I. Generate initial estimates of the biodistribution of the 64Cu-DOTA-pembrolizumab and the preferred dose of cold antibody.

II. Determine the dose of pre-administered unlabeled pembrolizumab that improves image quality by qualitative assessment by the radiologist of 64Cu-DOTA-pembrolizumab.

III. Evaluate the performance of 64Cu-DOTA-pembrolizumab in detecting tumor lesions.

OUTLINE: This is a dose-escalation study of 64Cu-DOTA-pembrolizumab.

Patients receive pembrolizumab intravenously (IV) over 30 minutes, and within 6 hours also receive 64Cu-DOTA-pembrolizumab via slow IV push over > 1 minute on day 0. Patients then undergo PET over 60 minutes on day 1.

After completion of study treatment, patients are followed up for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Ability to undergo standard PET imaging
* Plan to be treated with immunotherapy
* Karnofsky performance status (KPS) >= 50%
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 50/mm^3; platelet transfusions to help patients meet eligibility criteria are not allowed within 7 days before study enrollment
* Total bilirubin =< 1.5 x the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Calculated creatinine clearance >= 30 mL/min
* Woman of childbearing potential must be practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods; condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization; true abstinence (when this is in line with the preferred and usual lifestyle of the subject) during and after the study (6 months after the last dose of 64Cu-anti-PD1 [pembrolizumab]-N-hydroxysuccinimide [NHS]-DOTA for women)
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control, e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 6 months after receiving the last dose of study drug

Exclusion Criteria:

* Prior exposure to pembrolizumab or other anti-PD1 therapy
* Unable to tolerate PET scan
* Any condition that would, in the investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Female patients who are lactating or have a positive pregnancy test during the screening period
* Infection requiring systemic antibiotic therapy within 14 days prior to start of study treatment
* Subject is receiving concurrent chemotherapy or biologic or hormonal therapy for cancer treatment. Subject is receiving bone marrow stimulatory factors (e.g., granulocyte-macrophage colony-stimulating factor [GM-CSF]). Note: Concurrent use of hormones for noncancer-related conditions (e.g., insulin for diabetes) is acceptable
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Vaccination with live attenuated vaccines within 4 weeks of study agent administration
* Subject is currently using or has used immunosuppressive medication within 14 days prior to the study agent administration
* Intranasal, topical, inhaled, or local steroid injections (e.g., intra-articular injection)
* Chronic systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., infusion-related reactions, computed tomography [CT] scan premedication)
* Subject has plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary amyloidosis
* Subject has known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 < 50%
* Subject has known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, or their excipients
* Subject has history of primary immunodeficiency
* Subject is positive for human immunodeficiency virus (HIV-1), chronic or active hepatitis B, or active hepatitis A or C
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 3 days
  Toxicity will be graded according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events version 5.0. Observed toxicities will be summarized, for all dose levels, in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study agent(s) and reversibility or outcome.
Dose limiting toxicity | During the first 3 days post the administration of radiolabeled pembrolizumab

SECONDARY OUTCOMES:
Detection of lesions in the body by 64Cu-DOTA-pembrolizumab positron emission tomography | Up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Chaudhry, Principal Investigator — City of Hope Medical Center